CLINICAL TRIAL: NCT02744898
Title: A Phase 2 Feasibility Study of Abraxane and Carboplatin in Epithelial Neoplasms of the Uterus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-01156
Record Dates: First submitted 2016-04-15; First posted 2016-04-20 (Estimated); Results first posted 2020-03-18 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-08

CONDITIONS: Endometrial Cancer
Keywords: uterus; gynecological; corpus uteri
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Albumin-Bound Paclitaxel; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Carboplatin AUC and Abraxane 100mg/m2 (Experimental)
  Interventions: Drug: Carboplatin AUC; Drug: Abraxane

INTERVENTIONS:
Drug: Carboplatin AUC
Drug: Abraxane — 100mg/m2
  Other Names: Paclitaxel

SUMMARY:
The purpose of this study is to evaluate the safety of treatment with carboplatin and Abraxane in this patient population and determine the nature and degree of toxicities following treatment. The single stage open label Phase II feasibility study is designed to estimate the proportion of patients who can tolerate the proposed regimen for 6 cycles with no more than two dose level reductions.

ELIGIBILITY:
Inclusion Criteria:

* Female patients must have high risk resected stage I disease (papillary serous histology, clear cell histology or carcinosarcoma), advanced stage (III or IV, all histologies) or recurrent endometrial cancer (all histologies). Patients do not need measurable disease and can enroll following surgery.
* Patients may not have received prior cytotoxic chemotherapy. However, nonplatinum/non-taxane chemotherapy used for radiation sensitization is allowed. Patients may have received prior radiation therapy (including whole pelvic or vaginal brachytherapy), hormonal therapy, or therapy with biologic agents, but such therapy must be discontinued at least 2 weeks prior to entry on this study.
* If patients underwent surgery, and chemotherapy is indicated after surgery either as adjuvant or to treat residual disease, study treatment should be initiated within 8 weeks of surgery.
* In patients who have received prior radiation, at least 4 weeks should have elapsed since the completion of radiation therapy involving the whole pelvis or over 50% of the spine. If vaginal brachytherapy is planned with chemotherapy, it should be done before or after completion of chemotherapy treatment.
* Poorly differentiated histology, uterine papillary serous carcinoma, clear cell carcinoma or carcinosarcoma is acceptable as long as the predominant metastatic component is epithelial (versus sarcomatous).
* Patients may have synchronous endometrial and ovarian cancer primaries.
* Patients must have a GOG performance status of 0, 1, or 2
* Patients must be at least 18 years of age.
* Patients must understand and willingly sign an approved informed consent, and authorization permitting release of personal health information.
* Patients must have adequate liver function: AST and ALT ≤ 2.5 X upper limit of normal (ULN), and bilirubin ≤ 1.5mg/dL.
* Patients must have adequate bone marrow function: platelets ≥ 100,000 cells/mm3 (transfusion independent, defined as not receiving platelet transfusions within 7 days prior to laboratory sample), hemoglobin > 9.0g/dl and ANC ≥ 1,500 cells/mm3.
* Patients must have adequate renal function: creatinine < 1.5 mg/dL is recommended; however, institutional norms are acceptable.
* Patients must have < grade 2 pre-existing peripheral neuropathy (per CTCAE).

Exclusion Criteria:

* Other prior malignancies within 3 years, except non-melanoma skin cancers and synchronous ovarian primaries.
* Eligibility to a higher priority trial for first line or recurrent endometrial cancer (unless patient is unwilling to participate in such a trial).
* Patients with concomitant medical illness such as serious uncontrolled infection, or uncontrolled angina, which in the opinion of the treating physician, make the treatments prescribed on this study unreasonably hazardous for the patient.
* Patients who are pregnant or breastfeeding.
* Patients with third degree or complete heart block are not eligible unless a pacemaker is in place. Patients on medications, which alter cardiac conduction, such as digitalis, beta-blockers, or calcium channel blockers, or who have other conduction abnormalities or cardiac dysfunction could be entered at the discretion of the investigators.
* Patients with history of myocardial infarct within 6 months before enrollment, New York Heart Association (NYHA) class II or greater heart failure or symptoms suspicious for congestive heart failure are not eligible unless a LVEF in the past 6 months is documented to be 50% or greater. Patients who have had a LVEF (performed for any reason) that is less than 50% in the past 6 months are ineligible.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2018-08-17 (Actual); Study Completion 2020-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Franco Muggia, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Perlmutter Cancer Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Carboplatin AUC and Abraxane 100mg/m2: Carboplatin AUC
  Abraxane: 100mg/m2
Period: Overall Study
Arm/Group | Carboplatin AUC and Abraxane 100mg/m2
Started | 23
Completed | 19
Not Completed | 4
Not completed — Progressive Disease | 2
Not completed — Physician Decision | 1
Not completed — Toxicity | 1

BASELINE CHARACTERISTICS:
Population: 1-MD Decision
  1. Drug toxicity
  2. progressive disease
Groups:
- Carboplatin AUC and Abraxane 100mg/m2: Approximately 23 patients will be enrolled in this study at the Laura & Isaac Perlmutter Cancer Center at NYU Langone.There is a total of 17 study visits, including the screening visit to determine if you are eligible to participate. This study will be an out-patient study.
Arm/Group | Carboplatin AUC and Abraxane 100mg/m2
Number analyzed (Participants) | 23
Age, Continuous [Mean (Full Range); unit: years] | 65 [43 to 73]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 9
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: Tolerability Measured Completion of Dose Regimen
Description: Tolerability for an individual patient will be defined as remaining on the study for 6 cycles with two or fewer dose reductions.
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Carboplatin AUC and Abraxane 100mg/m2
Number analyzed (Participants) | 19
Participants | 16

2. Secondary Outcome: Progression-Free Survival (PFS) at Month 24
Description: PFS is defined as the time from first dosing to the first observation of disease progression or death due to any cause. PFS was estimated beyond the collected data using Kaplan Meier methods.
Time Frame: Up to Month 24
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Carboplatin AUC and Abraxane 100mg/m2
Number analyzed (Participants) | 23
Months | 28.2 [12.1 to NA] — Not releasable (NR); insufficient number of participants with events.

3. Secondary Outcome: Objective Response Rate (ORR) as Measured by RECIST 1.1 at Month 24
Description: ORR is the number of patients whose best tumor response outcome by Month 24 is a Complete Response (CR) or Partial Response (PR), divided by the total number of evaluable patients.
  Per the Response Evaluation Criteria in Solid Tumors (RECIST v1.1.):
  CR = Disappearance of all target lesions; PR = At least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD
Time Frame: Up to Month 24
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Carboplatin AUC and Abraxane 100mg/m2
Number analyzed (Participants) | 23
Percentage of participants | 33.3 [7.5 to 70.1]

ADVERSE EVENTS:
Time Frame: 24 Months
Arm/Group | Carboplatin AUC and Abraxane 100mg/m2
All-Cause Mortality (participants affected / at risk) | 0/23
Serious Adverse Events (participants affected / at risk) | 3/23
Other Adverse Events (participants affected / at risk) | 23/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carboplatin AUC and Abraxane 100mg/m2 (N=23)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Vomiting (General disorders) | 1 (1)
Dehydration (General disorders) | 1 (1)
Hypoalbuminemia (General disorders) | 1 (1)
Lymphocyte count decreased (Blood and lymphatic system disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Syncope (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Myalgia (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carboplatin AUC and Abraxane 100mg/m2 (N=23)
Abdominal Pain (Gastrointestinal disorders) | 4 (4)
Absolute Neutrophilous Count Decreased (Blood and lymphatic system disorders) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1)
Alanine Aminotransferase Increased (Renal and urinary disorders) | 5 (5)
Alkaline Phosphatase Elevated (Blood and lymphatic system disorders) | 1 (1)
Alkaline Phosphatase Increased (Blood and lymphatic system disorders) | 6 (6)
Allergic Reaction (General disorders) | 1 (1)
Alopecia (Congenital, familial and genetic disorders) | 16 (16)
Alt Increased (Blood and lymphatic system disorders) | 3 (3)
Anc Decreased (Blood and lymphatic system disorders) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 20 (20)
Anorexia (Psychiatric disorders) | 11 (11)
Anxiety (Psychiatric disorders) | 3 (3)
Arthralgia (Psychiatric disorders) | 3 (3)
Aspartate Aminotransferase Increased (Blood and lymphatic system disorders) | 7 (7)
Ast Increased (Blood and lymphatic system disorders) | 3 (3)
B/L Deep Vein Thrombosis (Cardiac disorders) | 1 (1)
B/L Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Back Pain (Injury, poisoning and procedural complications) | 1 (1)
Blood Bilirubin Increased (Blood and lymphatic system disorders) | 1 (1)
Body Aches(Myalgias) (General disorders) | 1 (1)
Chest Pain (General disorders) | 1 (1)
Colitis (Metabolism and nutrition disorders) | 1 (1)
Constipation (General disorders) | 11 (11)
Cough (General disorders) | 1 (1)
Cough/Clear Sputum (General disorders) | 1 (1)
Creatinine Increased (Hepatobiliary disorders) | 4 (4)
Decreased Anc (Blood and lymphatic system disorders) | 2 (2)
Decreased Neutrolphil Count (Blood and lymphatic system disorders) | 3 (3)
Decreased Platelet Count (Blood and lymphatic system disorders) | 3 (3)
Decreased Sodium (General disorders) | 1 (1)
Decreased White Blood Cell Count (Blood and lymphatic system disorders) | 6 (6)
Dehydration (General disorders) | 4 (4)
Diarrhea (General disorders) | 10 (10)
Dizziness (General disorders) | 4 (4)
Dry Skin (General disorders) | 1 (1)
Dyseusia (General disorders) | 1 (1)
Dysgeusia (General disorders) | 3 (3)
Dyspepsia (General disorders) | 1 (1)
Dyspnea (General disorders) | 2 (2)
Ear Infection (General disorders) | 0 (0)
Edema Limbs (General disorders) | 2 (2)
Elevated Alkaline Phosphatase (Blood and lymphatic system disorders) | 1 (1)
Elevated Alt (Blood and lymphatic system disorders) | 2 (2)
Elevated Creatinine (Blood and lymphatic system disorders) | 1 (1)
Elevated Potassium (Blood and lymphatic system disorders) | 2 (2)
Elevated Total Bilirubin (Blood and lymphatic system disorders) | 1 (1)
Epistaxis (General disorders) | 1 (1)
Eye Disorders (Eye disorders) | 1 (1)
Facial Flushing (General disorders) | 1 (1)
Fall (General disorders) | 1 (1)
Fatigue (General disorders) | 16 (16)
Flu Like Symptoms (General disorders) | 1 (1)
Gastroesophageal Reflux Disease 22 (General disorders) | 1 (1)
Generalized Weakness (General disorders) | 1 (1)
Gi Distress/Abdominal (General disorders) | 1 (1)
Gingival Pain (General disorders) | 1 (1)
Gum Infection (General disorders) | 1 (1)
Headache (General disorders) | 2 (2)
Hot Flashes (General disorders) | 1 (1)
Hypercalcemia (General disorders) | 1 (1)
Hyperkalemia (General disorders) | 1 (1)
Hypernatremia (General disorders) | 4 (4)
Hypertension (General disorders) | 1 (1)
Hypoalbuminemia (General disorders) | 1 (1)
Hypocalcemia (General disorders) | 1 (1)
Hypokalemia (General disorders) | 7 (7)
Hypomagnesemia (General disorders) | 2 (2)
Increased Alkaline Phospatase Level (General disorders) | 1 (1)
Increased Alkaline Phosphatase (General disorders) | 1 (1)
Injection Site Reaction (General disorders) | 1 (1)
Insomnia (General disorders) | 2 (2)
Intermittent Abdominal Pain (General disorders) | 1 (1)
Intermittent Anorexia (General disorders) | 1 (1)
Intermittent Blurred Vision (General disorders) | 1 (1)
Intermittent Decreased Platelets (General disorders) | 1 (1)
Intermittent Diarrhea (General disorders) | 1 (1)
Intermittent Dysgeusia (General disorders) | 1 (1)
Intermittent Fatigue (General disorders) | 2 (2)
Intermittent Hyperglycemia (General disorders) | 1 (1)
Intermittent Myalgias (General disorders) | 1 (1)
Intermittent Nausea (General disorders) | 7 (7)
L E Edema (General disorders) | 1 (1)
Le Edema (General disorders) | 1 (1)
Left Arm Pain (General disorders) | 1 (1)
Left Quadrant Pain (General disorders) | 1 (1)
Left-Hand Neuropathy (General disorders) | 1 (1)
Leukocytosis (General disorders) | 1 (1)
Leukopenia (General disorders) | 1 (1)
Low White Blood Cell Count (General disorders) | 1 (1)
Lymphocyte Count Decreased (General disorders) | 4 (4)
Memory Impairment (General disorders) | 1 (1)
Menorrhagia (General disorders) | 1 (1)
Mucositis Oral (General disorders) | 1 (1)
Muscle Weakness Upper Limb (General disorders) | 1 (1)
Musculoskeletal And Connective Tissue Disorder (General disorders) | 0 (0)
Musculoskeletal Pain (General disorders) | 1 (1)
Myalgia (General disorders) | 4 (4)
Nail Discoloration (General disorders) | 2 (2)
Nail Infection (General disorders) | 1 (1)
Nail Loss (General disorders) | 1 (1)
Nasal Congestion (General disorders) | 1 (1)
Nausea (General disorders) | 12 (12)
Neck Pain (General disorders) | 1 (1)
Neuotrophil Count Decreased (General disorders) | 1 (1)
Neuropathy (General disorders) | 1 (1)
Neutropenia (General disorders) | 1 (1)
Neutrophil Count Decreased (General disorders) | 8 (8)
Pain (General disorders) | 4 (4)
Pain (Tooth) (General disorders) | 1 (1)
Pain In Extremity (General disorders) | 1 (1)
Palpitations (General disorders) | 1 (1)
Paresthesia (General disorders) | 5 (5)
Pelvic Pain (General disorders) | 5 (5)
Peridontal Disease (General disorders) | 1 (1)
Peripheral Neuropathy (General disorders) | 2 (2)
Peripheral Sensory Neuropathy (General disorders) | 2 (2)
Photosensitivity (General disorders) | 1 (1)
Platelet Count (General disorders) | 1 (1)
Platelets Decresed (General disorders) | 3 (3)
Poor Venous Access (General disorders) | 0 (0)
Pruritis (General disorders) | 1 (1)
Rash Acneiform (General disorders) | 1 (1)
Renal And Urinary Disorders (Renal and urinary disorders) | 1 (1)
Right Leg Pain (General disorders) | 1 (1)
Scalp Rash (General disorders) | 1 (1)
Shortness Of Breath (General disorders) | 2 (2)
Skin And Subcutaneous Tissue Disorders (General disorders) | 1 (1)
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 (2)
Skin Infection (Skin and subcutaneous tissue disorders) | 1 (1)
Small Intestinal Obstruction (Infections and infestations) | 1 (1)
Syncope (General disorders) | 1 (1)
Tachycardia (General disorders) | 2 (2)
Thrombocytopenia (General disorders) | 3 (3)
Thromboembolic Event (General disorders) | 2 (2)
Toothache (General disorders) | 1 (1)
Total Bilirubin Elevated (General disorders) | 2 (2)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Urinary Frequency (General disorders) | 2 (2)
Urinary Urgency (General disorders) | 2 (2)
Vomiting (General disorders) | 3 (3)
Wbc Decreased (General disorders) | 1 (1)
Weight Loss (General disorders) | 1 (1)
White Blood Cells Decreased (General disorders) | 9 (9)
Wound Complication (General disorders) | 1 (23)
Right Leg Swelling (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-19): https://cdn.clinicaltrials.gov/large-docs/98/NCT02744898/Prot_SAP_000.pdf